CLINICAL TRIAL: NCT02687854
Title: Real-world Comparative Effectiveness of Apixaban Versus VKA
Brief Title: Real-world Comparative Effectiveness of Apixaban Versus Vitamin K Antagonist
Acronym: PIXI-F
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18731
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation (NVAF); Prevention; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — apixaban; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Apixaban: Non-valvular atrial fibrillation patients who were initiated on apixaban for stroke prevention
  Interventions: Drug: Apixaban
- Vitamin K antagonist: Non-valvular atrial fibrillation patients who were initiated on Vitamin K antagonist for stroke prevention
  Interventions: Drug: Vitamin K antagonist

INTERVENTIONS:
Drug: Apixaban — As prescribed by treating physicians
  Groups: Apixaban
Drug: Vitamin K antagonist — As prescribed by treating physicians
  Groups: Vitamin K antagonist

SUMMARY:
To obtain a better understanding on the comparative effectiveness of apixaban versus VKA (Vitamin K antagonist) for stroke prevention in patients with NVAF (Non-valvular atrial fibrillation) in a real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* NVAF will be defined as the occurrence of 2 or more inpatient or outpatient claims with ICD-9 427.31 as the diagnosis code at any time in the patient's data history prior to inclusion
* Patients will be required to have 180 days of enrollment for the assessment of baseline characteristics
* CHA2DS2-Vasc (C: Congestive heart failure; H: Hypertension; A2: Age ≥75 years; D: Diabetes mellitus; S2: prior Stroke or TIA or Thromboembolism; V: Vascular disease; A: Age 65-74 years; Sc: Sex category) score ≥2 during the 180 days prior to index apixaban use baseline period

Exclusion Criteria:

* Patients <18 years of age
* Patients with valvular AF (Atrial fibrillation)
* Pregnancy
* Malignant cancers
* Transient cause of AF
* Patients with VTE (Venous thromboembolism) (pulmonary embolism or DVT (Deep Vein Thrombosis))
* Patients with major surgery defined as hip or knee replacement
* Prescriptions of OACs (Oral anticoagulants) (apixaban, warfarin, dabigatran, rivaroxaban) before index date
* Prescription of more than one OAC on the index date
* Patient with any of the events defined in the composite endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation (NVAF)
Sampling Method: Non-Probability Sample
Enrollment: 18591 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Hospitalization Events (composite endpoint) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- New York, New York, United States